CLINICAL TRIAL: NCT04249388
Title: Rethink Pulmonary Rehabilitation (REPORT Study)
Brief Title: Characteristics of People With Advanced Chronic Obstructive Pulmonary Disease (COPD) - A Multicenter Study
Acronym: REPORT
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Hillerod Hospital, Denmark (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Henrik Hansen, Principal Investigator, Copenhagen University Hospital, Hvidovre
Other Study IDs: 19072886
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Decliners of Pulmonary Rehabilitation: No intervention, just observation
  Interventions: Other: No Intervention, just observation

INTERVENTIONS:
Other: No Intervention, just observation — No Intervention, just observation

SUMMARY:
Pulmonary rehabilitation (PR) is a cornerstone of care for people with COPD. There is robust evidence that PR improves exercise capacity, enhances health-related quality of life (QoL) and reduces healthcare utilization. PR is strongly recommended in guidelines for COPD management. Despite the compelling evidence for its benefits, PR is delivered to less than 30% of people with COPD. Access is particularly challenging, an especially for those with the most progressed disease stages.

We recently completed a randomized clinical trial, showing that approximately 1.100 patients annually are offered conventional hospital-based PR during routine consultations in the Capital Region of Denmark, but at least 700 patients declines participation.

No major cohort studies have been published from people with severe and advanced COPD who opt out of traditional pulmonary rehabilitation. By establishing such cohort study, objective and qualitative knowledge from assessments and patient interviews is collected in patients we have very limited access to and knowledge of. Additionally, the collected data will give a deeper insight and understanding and possibly enable us to design new delivery models to be tested in proper study designs.

DETAILED DESCRIPTION:
Objective This cohort study aims to describe and understand differences and similarities in characteristics among people with severe and advanced COPD who opt-in or opt out of PR services.

The study includes data from: socio-demographic, anthropometric, physical (function, activity, muscle strength, balance) characteristics as well as self-reported symptoms of anxiety, depression, fatigue, pain, lung symptoms, quality of life, sleep-quality, mortality, hospitaladmissions, length of stay and qualitative patient interviews.

Data from our completed trial study (NCT02667171) will be used as the opt-in PR comparison cohort.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD defined as a ratio of forced expiratory volume at one second (FEV1) to forced vital capacity < 0.70
* FEV1 <50%, corresponding to severe or very severe COPD
* Symptoms equivalent to the Medical Research Council (MRC) from 2 to 5
* Declines to participate in a conventional out-patient hospital-based PR program

Exclusion Criteria:

* Concurrent participation in or recent completion of pulmonary rehabilitation within the last twelve months.
* Dementia/ Cognitive impairment or uncontrolled psychiatric illness,
* An impaired hearing and / or vision which causes the instructions in the assessment is not understood.
* language difficulties which causes inability to follow instruction or complete patient reported outcome measures (PROM.)
* Any comorbidity that are contraindicated to the assesment protocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study of patients with COPD who declines participation in a conventional out-patient hospital-based PR program.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in points. Lower score indicates improvement

SECONDARY OUTCOMES:
6-Minute Walk Test Distance (6MWD) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes i meters. High is better
Hospital Anxiety and Depression Scale (HADS) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in point. Low score is better
Euro-Qol (EQ5D) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in Visual analogue scale (VAS). Higher VAS is better
Brief Pain Inventory (BPI) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in points. Low is better
Multidimensional Fatigue Inventory (MFI-20) | baseline and 52 weeks reassessment, (potentially 104 weeks reassesment)
  Observation of changes in points. Low is better
Short Physical Performance Battery (SPPB) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in point. High is better
Hand-Grip Strength (JAMAR) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in kilo. High is better
30 seconds sit-to-stand test (30sec-STS) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in repetitions. High is better
Pittsburgh Sleep Quality Index (PSQI) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in point. Low score is better
Number of hospital admissions (respiratory and all-cause) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in actual numbers. Low is better
Length of hospital admissions (respiratory and all-cause) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in days. Low is better
Out-patient visits | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in actual number. Low is better
Mortality (respiratory and all-cause) | baseline and 52 weeks reassessment, (potentially 104 weeks reassesment)
  Observation of changes as number of deaths. Low is better
Timed Up and Go Test | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment)
  Observation of changes in seconds. Low is better
Activity level (ActivPAL) | baseline and 52 weeks reassessment, (potentially 104 weeks reassessment) - Worn by the patients around the clock for 5 days
  Observation of changes in steps per day. High is better

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suppli Ulrik, MD, DMSc, Study Chair — Hvidovre University Hospital, Respiratory Department and Research Unit
Locations (4):
- Denmark (4):
  - Bispebjerg and Frederiksberg University Hospital, Copenhagen, Copenhagen North West
  - Amager and Hvidovre University Hospital, Hvidovre, Danmark
  - Gentofte and Herlev University Hospital, Gentofte Municipality, Hellerup
  - Nordsjaelland University Hospital, Hillerød

IPD SHARING:
Plan to Share IPD: Yes
Proposal for data use should be addressed to Henrik.hansen.09@regionh.dk
  Data access in Denmark are under very strict juristic data protection law.
  Any possible access or sharing demands a part application to
  1. Danish Data Protection Agency,
  2. Ethics Committee of the Capital Region
  3. National Health Data Authorities.
  Only if the applications are approved data will be considered available for sharing. The authors will not be able to support this process and a prolonged process must be expected.
Supporting Information: SAP, Analytic Code
Time Frame: unresolved
Access Criteria: Please read plan description